CLINICAL TRIAL: NCT03083912
Title: Effect of High Protein, High-calorie Nutritional Supplementation in Malnourished Elderly in Nursing Homes. A Prospective, Observational, Multicentric Study (PROT-e-GER Study)
Brief Title: Effect of High Protein, High-calorie Oral Nutritional Supplementation in Malnourished Elderly in Nursing Homes.
Acronym: PROT-e-GER
Status: Completed | Type: Observational
Sponsor: Hospital Viamed Valvanera, Spain (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Vincenzo Malafarina, MD MSc, MD, MSc, PhD3, University of Navarra
Other Study IDs: PROT-e-GER
Record Dates: First submitted 2016-10-25; First posted 2017-03-20 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Other Malnutrition
Keywords: Malnutrition; Disability; Oral Nutritional Supplementation
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fortimel Complete: All of the residents included receive ONS
  Interventions: Dietary Supplement: Fortimel Complete

INTERVENTIONS:
Dietary Supplement: Fortimel Complete — The residents included receive 2 bottle por day.
  Other Names: ONS

SUMMARY:
The hypothesis of this study is that the administration of a high-calorie high-protein oral nutritional supplement twice a day for three months to elderly malnourished in residents in Spain is associated with improved nutritional status, with an increase in body weight of between 5 and 8%, and an improvement in functional status, with low incidence of complication.

DETAILED DESCRIPTION:
A prospective, multi centric, observational study. The study is conducted in elderly living in nursing homes in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65 years,
* Living in nursing homes,
* Malnutrition treated with an hyper-caloric oral nutritional supplementation (1.3 Kcal / ml) and high-protein (protein 20%).

Exclusion Criteria:

* Tube feeding (nasogastric or gastrostomy)
* Terminally ill or palliative treatment and residents with life expectancy of less than 6 months
* Special nutritional requirements (for example by intestinal malabsorption, short bowel residents or specific nutrition for renal insufficiency).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Malnourished elderly living in nursing homes
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Improve weight | 3 months
  Difference between the weight of the residents at the beginning and at the end of the study

SECONDARY OUTCOMES:
SPPB scale | 3 months
  Functional status at the end of the study
Barthel index | 3 months
  Ability in Activities of Daily Living at the end of the study

OTHER OUTCOMES:
Number of drinking bottles during the study. | 3 months
  Evaluate the compliance with the oral nutritional supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Fernandez Bodas, Study Chair — Nutricia, Inc.; Alfonso Cruz Jentoft, MD PhD, Study Director — Head of Geriatric Department, Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malafarina V, Uriz-Otano F, Gil-Guerrero L, Iniesta R. The anorexia of ageing: physiopathology, prevalence, associated comorbidity and mortality. A systematic review. Maturitas. 2013 Apr;74(4):293-302. doi: 10.1016/j.maturitas.2013.01.016. Epub 2013 Feb 13. PMID 23415063
- [Background] van Nie-Visser NC, Meijers J, Schols J, Lohrmann C, Bartholomeyczik S, Spreeuwenberg M, Halfens R. Which characteristics of nursing home residents influence differences in malnutrition prevalence? An international comparison of The Netherlands, Germany and Austria. Br J Nutr. 2014 Mar 28;111(6):1129-36. doi: 10.1017/S0007114513003541. Epub 2013 Nov 18. PMID 24246053
- [Background] Salva A, Serra-Rexach JA, Artaza I, Formiga F, Rojano I Luque X, Cuesta F, Lopez-Soto A, Masanes F, Ruiz D, Cruz-Jentoft AJ. [Prevalence of sarcopenia in Spanish nursing homes: Comparison of the results of the ELLI study with other populations]. Rev Esp Geriatr Gerontol. 2016 Sep-Oct;51(5):260-4. doi: 10.1016/j.regg.2016.02.004. Epub 2016 Apr 9. Spanish. PMID 27068239
- [Background] Camina-Martin MA, de Mateo-Silleras B, Malafarina V, Lopez-Mongil R, Nino-Martin V, Lopez-Trigo JA, Redondo-del-Rio MP. Nutritional status assessment in geriatrics: Consensus declaration by the Spanish Society of Geriatrics and Gerontology Nutrition Work Group. Maturitas. 2015 Jul;81(3):414-9. doi: 10.1016/j.maturitas.2015.04.018. Epub 2015 May 14. PMID 26025067
- [Background] Malafarina V, Uriz-Otano F, Iniesta R, Gil-Guerrero L. Effectiveness of nutritional supplementation on muscle mass in treatment of sarcopenia in old age: a systematic review. J Am Med Dir Assoc. 2013 Jan;14(1):10-7. doi: 10.1016/j.jamda.2012.08.001. Epub 2012 Sep 13. PMID 22980996
- [Background] Lozano-Montoya I, Velez-Diaz-Pallares M, Abraha I, Cherubini A, Soiza RL, O'Mahony D, Montero-Errasquin B, Correa-Perez A, Cruz-Jentoft AJ. Nonpharmacologic Interventions to Prevent Pressure Ulcers in Older Patients: An Overview of Systematic Reviews (The Software ENgine for the Assessment and optimization of drug and non-drug Therapy in Older peRsons [SENATOR] Definition of Optimal Evidence-Based Non-drug Therapies in Older People [ONTOP] Series). J Am Med Dir Assoc. 2016 Apr 1;17(4):370.e1-10. doi: 10.1016/j.jamda.2015.12.091. Epub 2016 Feb 5. PMID 26857298